CLINICAL TRIAL: NCT07265869
Title: A Placebo-controlled, Randomized, Double-masked, Cross-over Acute Intervention Study Investigating the Effects of Cocoa Flavanols on Peripheral Endothelial Function in the Context of Prolonged Sitting in Healthy Older Adults
Brief Title: Can Cocoa Flavanols Protect Endothelial Function During Prolonged Sitting in Healthy Older Adults?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: ERN_19-0851B
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Ageing
Keywords: vascular function; endothelial function; flow-mediated dilatation; flavanols; cocoa; flavonoids; polyphenols; sitting; sedentary; ageing; older adults; functional Near-Infrared Spectroscopy
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flavanol cocoa powder (Experimental): 12 g of fat-reduced natural cocoa powder containing 695 mg of total flavanols, including 150 mg (-)-epicatechin
  Interventions: Dietary Supplement: High-flavanol cocoa powder
- Low-flavanol cocoa powder (Placebo Comparator): 12 g of fat-reduced alkalized cocoa powder containing 5.6 mg of total flavanols
  Interventions: Dietary Supplement: Low-flavanol cocoa powder

INTERVENTIONS:
Dietary Supplement: High-flavanol cocoa powder — 12 g of a fat-reduced natural cocoa powder containing 150 mg of (-)-epicatechin, and 695 mg of total flavanols
  Arms: High-flavanol cocoa powder
Dietary Supplement: Low-flavanol cocoa powder — 12 g of a fat-reduced alkalized cocoa powder containing 5.6 mg of total flavanols
  Arms: Low-flavanol cocoa powder

SUMMARY:
Sitting time is high in older adults and has been shown to temporarily impair endothelial function and blood pressure. Flavanols, plant-derived compounds, acutely enhance endothelial function and reduce Blood pressure in older adults. The aim of this study is to investigate whether acute ingestion of cocoa flavanols can improve peripheral endothelial function and blood pressure during prolonged sitting in healthy older adults.

In a randomised, double-blinded, cross-over, placebo-controlled human study, 20 healthy older adults will consume either a high-flavanol (695 mg) or low-flavanol (5.6 mg) cocoa beverage immediately before a 2-hour sitting bout. Flow-mediated dilation (FMD) of the superficial femoral (SFA; primary outcome) and brachial (BA) arteries, and blood pressure, were assessed before and after sitting. Microvasculature haemodynamics were assessed in the gastrocnemius before, during, and after sitting. It is hypothesized that the high flavanol cocoa will prevent declines in brachial and superficial femoral Flow-mediated dilatation post sitting.

DETAILED DESCRIPTION:
Older individuals are estimated to spend more than 10 hours in their waking day in sedentary activities , which can include sitting bouts lasting up to 5.4 hours/day . Greater sedentary time was found to be associated with a significantly increased risk of cardiovascular diseases and all-cause mortality. Several experimental studies have shown that even just one isolated episode of prolonged sitting (from 1 to 6 hours) has detrimental effects on human endothelial function, as measured by flow-mediated dilation (FMD).

Flavonoid-rich foods are typically consumed in high amounts in cardioprotective diets, with evidence from both observational and Randomised Controlled Trials showing flavonoids to improve biomarkers of cardiovascular health. Flavanols, a sub-group of flavonoids present in unprocessed cocoa, have been extensively shown to act quickly within the vasculature, improving both brachial Flow-mediated dilatation and lower-limb common femoral artery (CFA) Flow-mediated dilatation within 2 hours of intake in older adults.

The aim of the current study is to examine whether acute consumption of cocoa flavanols prior to a 2-hour bout of uninterrupted sitting can be beneficial in improving endothelial function (as measured by Flow mediated dilatation) in the upper-limb Brachial Artery (BA) and lower-limb Superficial Femoral Artery (SFA) in older adults, as well as downstream, muscle microvascular function. We will further investigate whether cocoa flavanols can prevent sitting-induced increases in blood pressure in older adults. We hypothesise that cocoa flavanols would be effective at rescuing upper- and lower-limb Flow-mediated dilatation and improve blood pressure during uninterrupted sitting in older age

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* aged 65 or more

Exclusion Criteria:

* history or symptoms of cardiovascular, renal, pulmonary, metabolic, or neurologic disease, hypertension (blood pressure higher than 140/90 mm Hg, based on recent guidelines), diabetes mellitus, anaemia, asthma, immune conditions, or high cholesterol.
* smoker
* individuals who were on weight-reducing diets
* individuals taking anticoagulants,
* had recently undergone prolonged bed-rest periods
* have been on antibiotics in the previous 3 months
* have an infection at present (e.g. cold) or viral infection

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation of the superficial femoral artery | Change from pre-intervention baseline to 2 hours post intervention /2 hours post sitting
  Flow-mediated dilatation (FMD) of the superficial femoral artery. Expressed as percent FMD: change in brachial diameter from baseline to peak dilation following 5 minutes of arterial occlusion. Brachial artery diameter and blood flow will be measured using Doppler ultrasonography (uSmart 3300, Terason).

SECONDARY OUTCOMES:
Flow-mediated dilatation of the brachial artery | Change from pre-intervention baseline to 2 hours post-intervention/ 2hours post sitting
  Flow-mediated dilatation (FMD) of the brachial artery. Expressed as percent FMD: change in brachial diameter from baseline to peak dilation following 5 minutes of arterial occlusion. Brachial artery diameter and blood flow will be measured using Doppler ultrasonography (uSmart 3300, Terason).
Tissue oxygenation index (TOI) of Gastrocnemius skeletal muscle | Change from pre-intervention baseline to 2 hours post-intervention / 2 hours of sitting
  Tissue Oxygenation Index (percent TOI) will be assessed by functional Near-Infrared Spectroscopy (fNIRS) on the medial head of the gastrocnemius muscle during 5 min of superficial femoral arterial occlusion and 5 min of post-occlusion (reactive hyperaemia). The NIRS device measures changes in chromophore concentrations of oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb), providing depth-resolved measures of total tissue oxygen saturation.
Normalized haemoglobin index (nTHI) of the gastrocnemius skeletal muscle | Change from pre-intervention baseline to 2 hours post-intervention/2 hours sitting
  Normalized haemoglobin index (relative value of total haemoglobin normalised to the initial value, nTHI) content (a.u.) will be assessed by functional Near-Infrared Spectroscopy (fNIRS) on the medial head of the gastrocnemius muscle during 5 minutes of superficial femoral arterial occlusion and 5 minutes of post-occlusion (reactive hyperaemia).
Tissue oxygenation index (TOI) of Gastrocnemius skeletal muscle during 2 hours of sitting | Post-intervention time points considered during sitting were 0 , 10 , 60 and 120 minutes.
  Tissue Oxygenation Index (percent TOI) will be assessed by functional Near-Infrared Spectroscopy (fNIRS) on the medial head of the gastrocnemius muscle continuously during 2 hours of sitting. The NIRS device measures changes in chromophore concentrations of oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb), providing depth-resolved measures of total tissue oxygen saturation. Post-intervention time points considered during sitting were 0 minutes , 10 minutes, 60 minutes, and 120 minutes. For each time point, data were averaged over a 60-second period.
Normalized haemoglobin index (nTHI) of Gastrocnemius skeletal muscle during 2 hours of sitting | Post-intervention time points considered during sitting were 0 min , 10 min, 60 min and 120 min.
  Normalized haemoglobin index (relative value of total haemoglobin normalised to the initial value, nTHI) content (a.u.) will be assessed by functional Near-Infrared Spectroscopy (fNIRS) on the medial head of the gastrocnemius muscle continuously during 2 hours of sitting. Post-intervention time points considered during sitting were 0 min , 10 min, 60 min, and 120 min. For each time point, data were averaged over a 60-second period.
Brachial Systolic Blood Pressure (SBP) | Change from pre-intervention baseline to 2 hours post-intervention / 2 hours of sitting
  Resting systolic blood pressure (mmHg) will be measured using an automated oscillometric blood pressure monitor, with a cuff attached to the right upper arm, following at least 10 minutes rest.
Brachial Diastolic Blood Pressure (DBP) | Change from pre-intervention baseline to 2 hours post-intervention / 2 hours of sitting
  Resting diastolic blood pressure (mmHg) will be measured using an automated oscillometric blood pressure monitor, with a cuff attached to the right upper arm, following at least 10 minutes rest.
Heart Rate | Change from pre-intervention baseline to 2 hours post-intervention/2 hours sitting
  Resting Heart Rate (beats per minute) will be measured using an automated oscillometric blood pressure monitor, with a cuff attached to the right upper arm, following at least 10 minutes rest.
Resting Superficial Femoral Artery Blood Flow | Change from pre-intervention baseline to 2 hours post-intervention/2 hours sitting
  Superficial Femoral Artery Blood Flow velocity (ml min-1) will be measured using Doppler ultrasonography (uSmart 3300, Terason) interfaced with the Quipu analysis software. Superficial femoral artery blood flow is calculated using Superficial femoral artery blood velocity and diameter during 1 minute of recording in a resting state
Resting Brachial Artery Blood Flow | Change from pre-intervention baseline to 2 hours post-intervention/2 hours sitting
  Resting Brachial Artery Blood Flow velocity (ml min-1) will be measured using Doppler ultrasonography (uSmart 3300, Terason) interfaced with the Quipu analysis software. Brachial Artery blood flow is calculated using brachial artery blood velocity and diameter during1 minute of recording in a resting state
Superficial Femoral Artery Shear Rate | Change from pre-intervention baseline to 2 hours post-intervention/2 hours sitting
  Superficial Femoral Artery Shear Rate shear rate (s-1) will be measured using Doppler ultrasonography (uSmart 3300, Terason) interfaced with the Quipu analysis software, during 1 minute in the resting state
Brachial Artery Shear Rate | Change from pre-intervention baseline to 2 hours post-intervention/2 hours sitting
  Brachial Artery Shear Rate shear rate (s-1) will be measured using Doppler ultrasonography (uSmart 3300, Terason) interfaced with the Quipu analysis software, during 1 minute in the resting state

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport, Exercise & Rehabilitation Sciences, University of Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT07265869/ICF_000.pdf